CLINICAL TRIAL: NCT03305055
Title: Evaluating the Safety, Efficacy and Opiate Sparing Effects of Low-Dose, Slow Infusion Ketamine as a Battlefield Analgesic for Acute Pain in Burn Wounds.
Brief Title: RCT: Fentanyl Plus Ketamine Versus Fentanyl Alone for Acute Burn Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding withdrawn - slow enrollment
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00089761; NTI-NTRR15-13 (Other Grant/Funding Number: National Trauma Institute; Departement of Defense)
Record Dates: First submitted 2017-06-12; First posted 2017-10-09 (Actual); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Acute Pain; Wound Care; Posttraumatic Stress Disorder
Keywords: opioid; ketamine
MeSH Terms: conditions — Acute Pain; Stress Disorders, Post-Traumatic | interventions — Ketamine; Fentanyl; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, repeated exposure (twice daily, 7 days), safety and efficacy trial of Usual Care (fentanyl PLUS saline / placebo) versus Usual Care plus Study Drug Augmentation (fentanyl PLUS ketamine) in reducing acute pain severity assessed before, during and after wound care for acute burn injury in the Burn Center of an Academic Medical Center.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacy receives order from provider and then prepares the study drug in an unmarked, nondescript delivery system ("bag") and the study drug information is entered from the bag into the pump so that delivery that is timed and volume controlled per study protocol. This is hung next to patient, connected and started. Masked personnel include provider (order study drug protocol), nurse (wound care), data assessor (Research Assistant), and consenting participant (patient with acute burn).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fentanyl Plus Ketamine (Experimental): Study drug group
  1. Ketamine Loading Dose (Low Dose, Slow Infusion) =
     • 0.3 mg/kg; Initiated approximately 10 minutes before wound care start, pump set to deliver slowly over approximately 5 minutes, … Then,
  2. Fentanyl Loading Dose (UC, injection) =
     • 1 mcg / kg. This is given to participants in both Group 1 and Group 2 initiated < 1 minute prior to wound care.
  3. Ketamine (Study Drug, Infusion) = • 2.5 mcg/kg/min, Pump initiates infusion immediately after the fentanyl Loading Dose and continued for session duration. The nurse determines session end, then turns off infusion.
  Fentanyl PRN dose* = 1 mcg / kg. Provided when participant requires additional pain medication.
  Interventions: Drug: ketamine; Drug: Fentanyl
- Fentanyl Plus Saline (Active Comparator): Usual care group
  1. Saline Loading Dose (Low Dose, Slow Infusion) =
     • An identical volume of saline as that in 0.3 mg/kg of ketamine. Initiated approximately 10 minutes before wound care start, pump set to deliver slowly over approximately 5 minutes, (i.e., same time/rate as STUDY DRUG GROUP receives ketamine loading dose), … Then, ...
  2. Fentanyl Loading Dose (UC, injection) =
     • 1 mcg / kg: This is given to participants in both Group 1 and Group 2 initiated <1 minute prior to wound care.
  3. Saline (Placebo, Infusion) = • Identical volume of fluid as that in 2.5 mcg/kg/min of ketamine; Pump initiates infusion immediately after the fentanyl Loading Dose and continued for session duration. The nurse determines session end, then turns off infusion.
  FENTANYL PRN DOSE = 1 mcg / kg. Provided when participant requires additional pain medication.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: ketamine — Information included in arm descriptions
  Other Names: STUDY DRUG GROUP (Fentanyl plus Ketamine)
  Arms: Fentanyl Plus Ketamine
Drug: Fentanyl — Information included in arm descriptions
  Other Names: USUAL CARE GROUP (Fentanyl plus saline/placebo)

SUMMARY:
The Ketamine for Acute Pain in Burns study is a randomized, double-blind, parallel group trial (RCT) with active control (usual care) contrasting the efficacy and safety of "Ketamine Plus Opiate-based usual care" (O+K) with the safety and efficacy of the "Current Standard of Care". THe current standard of care is an opiate medication alone, Fentanyl (Usual Care-Opiate (UC-O), dose/timing as per Burn Center protocol).

DETAILED DESCRIPTION:
Department of Defense (DoD) and the U.S. Army Medical Research and Materiel Command (USAMRMC) are funding this RCT for the following reasons:

Primary Aims:

1. To evaluate the safety and efficacy of fentanyl (usual care) + placebo versus fentanyl + ketamine (low-dose, sub-anesthetic, slow-infusion) during twice daily burn wound care across a 7-day study period and 30 day outcome period.
2. To evaluate the opiate sparing effect of fentanyl (usual care) + placebo versus fentanyl + ketamine (low-dose, sub-anesthetic, slow-infusion) during the 7-day study period and 30 day outcome period.

and

Secondary Aims:

1. To determine the short and long term effect of the Ketamine Augmentation Condition versus the Usual Care Condition on symptoms and syndromes of posttraumatic stress disorder and of depression,
2. To evaluate several established and hypothesized moderators of the relationship between the Ketamine Augmentation Condition versus the Usual Care Condition on: 1) pain severity reported during wound care, 2) opiate use during wound care, 3) posttraumatic stress and 4) depression.

ELIGIBILITY:
Inclusion Criteria:

* Total Body Surface Area (TBSA) greater than or equal to 2%; Less than or equal to 40% TBSA
* English speaking
* pain in emergency room during initial wound evaluation (on admission) greater than 5 /10
* estimated length of stay greater than or equal to 5 days

Exclusion Criteria:

* requiring endotracheal intubation and sedation,
* severe hearing impairment,
* cognitive impairment status - Mini-Mental State Examination (MMSE) </=20,
* diminished capacity unable to provide informed consent;
* Past Medical History (PMH): insensate (eg. spinal cord injury, peripheral neuropathy)
* Safety: contraindication (e.g., potential drug interactions or medical comorbidities)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-16 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Fauerbach, PhD, Principal Investigator — Johns Hopkins University SOM; Kevin Gerold, DOJD, Principal Investigator — Johns Hopkins University SOM; Julie Caffrey, DO, Study Director — Johns Hopkins University SOM
Locations (1):
- Johns Hopkins Burn Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan not operationalized as yet.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available by 1 year after final data publication and remain available for indefinitely.
Access Criteria: Written request from faculty investigator to PI or Study Director specifying planned safety & monitoring plan and data analytic aims and hypotheses

RESULTS

PARTICIPANT FLOW:
Groups:
- Fentanyl Plus Ketamine: Study drug group
  1. Ketamine Loading Dose (Low Dose, Slow Infusion) =
     • 0.3 mg/kg; Initiated approximately 10 minutes before wound care start, pump set to deliver slowly over approximately 5 minutes, … Then,
  2. Fentanyl Loading Dose (UC, injection) =
     • 1 mcg / kg. This is given to participants in both Group 1 and Group 2 initiated < 1 minute prior to wound care.
  3. Ketamine (Study Drug, Infusion) = • 2.5 mcg/kg/min, Pump initiates infusion immediately after the fentanyl Loading Dose and continued for session duration. The nurse determines session end, then turns off infusion.
  Fentanyl PRN dose* = 1 mcg / kg. Provided when participant requires additional pain medication.
  ketamine: Information included in arm descriptions
  Fentanyl: Information included in arm descriptions
- Fentanyl Plus Saline: Usual care group
  1. Saline Loading Dose (Low Dose, Slow Infusion) =
     • An identical volume of saline as that in 0.3 mg/kg of ketamine. Initiated approximately 10 minutes before wound care start, pump set to deliver slowly over approximately 5 minutes, (i.e., same time/rate as STUDY DRUG GROUP receives ketamine loading dose), … Then, ...
  2. Fentanyl Loading Dose (UC, injection) =
     • 1 mcg / kg: This is given to participants in both Group 1 and Group 2 initiated <1 minute prior to wound care.
  3. Saline (Placebo, Infusion) = • Identical volume of fluid as that in 2.5 mcg/kg/min of ketamine; Pump initiates infusion immediately after the fentanyl Loading Dose and continued for session duration. The nurse determines session end, then turns off infusion.
  FENTANYL PRN DOSE = 1 mcg / kg. Provided when participant requires additional pain medication.
  Fentanyl: Information included in arm descriptions
Period: Overall Study
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Started | 2 | 2
Completed | 1 | 0
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (35.4) | 37 (15.6) | 40.5 (22.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Wound Care Pain
Description: Average Pain across 14 sessions between the 2 groups and related outcome measures up to 40 days following study enrollment.
Time Frame: Up to 40 days
Population: Data was not collected for the minimum threshold [per the statistical analysis plan] of 6-11 consecutive wound care sessions to assess this outcome measure
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Trajectory of Mean Wound Care Session Pain Within Sessions
Description: Trajectory of average pain within session
Time Frame: 7-days, within session
Population: as for outcome 1
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Trajectory of Mean Wound Care Session Pain Across Sessions
Description: Trajectory of average pain across 7 day study protocol
Time Frame: 7-Days across sessions
Population: as for outcome 1
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Opiate Sparing Effect
Description: Pro Re Nata (PRN) pain management or adjunct expressed in opiate equivalents (e.g., anxiolytic) or premed (e.g., non-protocol medications for pain, anxiety, etc); post-session (1 and 6 hours post session , e.g., pain, anxiolytic, etc).
Time Frame: 37 days
Population: Data was not collected for this outcome measure.
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Post Traumatic Stress Disorder (PTSD) Symptoms as Assessed by Davidson Trauma Scale
Description: PTSD symptoms score as assessed by Davidson Trauma Scale consisting of 17 items (symptoms) with each item measured for severity and frequency. Each item is rated 0 - 4. Overall score ranges from 0 to 136, with higher scores indicating higher frequency and severity.
Time Frame: 37 days
Population: as for outcome 1
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Depression Symptoms as Assessed by the Patient Health Questionnaire
Description: Severity and trajectory of depression symptoms as assessed by the Patient Health Questionnaire (PHQ) 9. The questionnaire has 9 items with each rated from 0 to 3. Overall scores ranges from 0 to 27 with 1-4 being minimal depression, 5-9 being mild depression, 10-14 being moderate depression, 15-19 being moderately severe depression and 20-27 being severe depression.
Time Frame: 37 days
Population: as for outcome 1
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: End of study (approximately 37 days)
Arm/Group | Fentanyl Plus Ketamine | Fentanyl Plus Saline
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fentanyl Plus Ketamine (N=2) | Fentanyl Plus Saline (N=2)
Pain at wound site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT03305055/Prot_SAP_000.pdf